CLINICAL TRIAL: NCT00948428
Title: A Multicenter, Double-Blind, Randomized, Parallel Group, Vehicle-Controlled Study to Determine the Clinical Equivalence of a Generic Imiquimod Cream, 5% and Aldara™ Cream in Subjects With Actinic Keratosis
Brief Title: Bioequivalence of Generic Imiquimod Cream, 5% When Compared to Aldara™ (Imiquimod) Cream, 5% in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D94-3101-07
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; imiquimod; therapeutic equivalence; bioequivalence
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Generic Imiquimod (Active Comparator): imiquimod cream, 5%
  Interventions: Drug: imiquimod
- Aldara™ (Active Comparator): Aldara™ (imiquimod) cream, 5%
  Interventions: Drug: Aldara™
- Vehicle cream (Placebo Comparator): Vehicle cream (Actavis)
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: imiquimod — 5% topical cream dispensed in individual 0.25 g sachets applied twice a week for 16 weeks
  Arms: Generic Imiquimod
Drug: Aldara™ — 5% topical cream dispensed in individual 0.25 g sachets applied twice a week for 16 weeks
  Arms: Aldara™
Drug: Vehicle Cream — Topical cream vehicle matching Generic imiquimod dispensed in individual 0.25 g sachets applied twice a week for 16 weeks
  Arms: Vehicle cream

SUMMARY:
At the end of the study, safety and efficacy outcome measures will be compared to determine a) if dosing with Generic Imiquimod cream, 5% is therapeutically equivalent to the currently marketed Aldara (imiquimod) cream, 5% and b) if both imiquimod 5% creams are superior in comparison to the Vehicle cream.

DETAILED DESCRIPTION:
A nationwide, multicenter, double-blind, vehicle-controlled parallel group comparison study of a Generic Imiquimod cream, 5% (Actavis Mid-Atlantic LLC) and currently marketed Aldara (imiquimod) cream, 5% (distributed by Graceway Pharmaceuticals, LLC) was conducted in subjects with actinic keratoses (AKs) on the face and/or anterior scalp in order to evaluate the therapeutic equivalence of these two active treatments and to establish superiority of the efficacy of these two products over a Vehicle cream. Subjects were randomized to one of three treatment groups on a 2:2:1 basis as follows: (1) Generic Imiquimod cream, 5%, (2) Aldara (imiquimod) cream, 5%, and (3) Vehicle cream. The duration of treatment was 16 weeks (± 7 days).

The primary efficacy endpoint was the proportion of subjects in each treatment group with Complete Clearance (having no clinically visible actinic keratosis lesions in the 25 cm2 contiguous treatment area at the 8-week post-treatment visit) of AK lesions. The secondary efficacy endpoints were the Partial Clearance rates, defined as the proportion of subjects with at least a 75% reduction in the number of AK lesions counted at Baseline at the end-of-treatment visit (Week 16, EOT) and at the 8 weeks post-treatment visit/test-of-cure (Week 24, TOC), and the proportion of subjects with Complete Clearance of AK lesions at the end-of-treatment (Week 16, EOT) visit.

A 90% Wald's confidence interval with Yate's continuity correction was constructed around the difference between the proportions of subjects with Complete Clearance of AK lesions in the active treatments (Generic Imiquimod minus Aldara) to evaluate therapeutic equivalence in the primary efficacy analyses. Two-sided, continuity-corrected statistics were used to evaluate the superiority of each active treatment's Complete Clearance rate over that of the Vehicle treatment. The therapeutic comparability evaluations in the per-protocol (PP) population were considered primary while those in the intent-to-treat (ITT) population were considered supportive. The superiority comparisons in the ITT population were considered primary while those in the PP population were considered supportive. If the 90% confidence interval (CI) around the difference between the Generic Imiquimod and Aldara Complete Clearance rates in the PP population were contained within the interval 0.20 to +0.20, and each of these rates was greater than, and statistically different (p<0.05) from, the Vehicle rate in the ITT population, then Generic Imiquimod and Aldara were considered to be therapeutically equivalent.

Secondary efficacy analyses were conducted on the proportion of subjects in each treatment group with Complete Clearance of AK lesions at the Week 16, EOT visit as well as evaluation of the Partial Clearance of AK lesions at both the EOT and TOC visits. The results at both the EOT visit (Week 16) and those at 8 weeks post-treatment (Week 24, TOC) were statistically analyzed by the same methods described for the primary efficacy variable.

Both EOT and TOC analyses were conducted in the ITT population. The TOC analysis was conducted in the PP population and the EOT analysis was conducted in the EOT PP population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were male or non-pregnant females, 18 years of age or older, in generally good health. Females who were post-menopausal, surgically sterile or using a medically acceptable form of birth control with a negative urine pregnancy test at the Baseline visit.
* Subjects provided written and verbal informed consent.
* Subjects presented to the clinic with at least 4 but no more than 12 visible, discrete nonhyperkeratotic, nonhypertrophic actinic keratosis lesions within a 25 cm2 Treatment Area on the face and/or anterior scalp.
* Subjects were willing and able to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

* Subjects who were lactating, or planning to become pregnant during the study.
* Subjects had hyperkeratotic, hypertrophic or large mat-like AKs within the 25 cm2 Treatment Area.
* Subjects who had the need or were planning to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Subjects who were immunosuppressed (e.g., HIV, systemic malignancy, graft vs. host disease, etc.).
* Subjects who experienced an unsuccessful outcome from previous imiquimod therapy.
* Subjects with known hypersensitivity or previous allergic reaction to any of the active or inactive components of the study drugs.
* Within 2 months: Facial and/or Anterior Scalp: laser resurfacing, photodynamic therapy, chemical peels, dermabrasion, topical application of 5-FU, imiquimod, diclofenac sodium or other treatments for AK or photodamage.
* Subjects who used the following systemic, oral or topical therapies for the periods specified prior to entry into the study:

Within 2 days: Topicals of any kind to the selected Treatment Area. Within 2 weeks: Facial topical medications: corticosteroids, alpha- hydroxyacids (e.g., glycolic acid, lactic acid, etc. greater than 5%), beta-hydroxyacid (salicylic acid greater than 2%), urea - greater than 5% or prescription retinoids (e.g., tazarotene, adapalene, tretinoin) to the face and/or anterior scalp.

Within 2 weeks: Cryotherapy to lesions adjacent to or within the 25 cm2 Treatment Area.

Within 4 weeks: Systemic steroid therapy: chemotherapeutic agents, psoralens, immunotherapy, or retinoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M. Winslow, Ph.D., Study Director — Actavis Mid-Atlantic LLC
Locations (20):
- United States (20):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Associates in Research, Inc., Fresno, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - FXM Research Corp., Miami, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Mt. Sinai School of Medicine, New York, New York
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - Rhode Island Hospital, Dermatopharmacology Division, Providence, Rhode Island
  - Dermatology Associates of Knoxville, P.C., Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce & Associates, P.A., Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream
Started | 185 | 185 | 92
Completed | 167 | 167 | 84
Not Completed | 18 | 18 | 8
Not completed — Withdrawal by Subject | 6 | 12 | 7
Not completed — Adverse Event | 6 | 3 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Intercurrent Illness | 1 | 0 | 0
Not completed — Non-compliance | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Using Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream | Total
Number analyzed (Participants) | 181 | 179 | 89 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (10.1) | 66.7 (10.4) | 66.7 (9.9) | 66.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 20 | 13 | 62
  Male | 152 | 159 | 76 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 2 | 13
  Not Hispanic or Latino | 176 | 173 | 87 | 436
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 181 | 179 | 89 | 449
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Each Treatment Group With Complete Clearance of AK Lesions at the Test of Cure Visit (Week 24)
Time Frame: Week 24
Population: Using Per-Protocol Population (PP)
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream
Number analyzed (Participants) | 158 | 151 | 76
Participants | 74 | 72 | 7
Statistical Analysis 1: Comparison: Generic Imiquimod vs Aldara™; Test type: Equivalence — If the 90% confidence interval around the difference between the Generic Imiquimod and Aldara Complete Clearance rates in the PP population were contained within the interval -0.20 to +0.20, and each of these rates was greater than, and statistically different (p<0.05) from, the Vehicle rate in the ITT population, then Generic Imiquimod and Aldara were considered to be therapeutically equivalent; Mean Difference (Net) = -0.85, 90% CI 2-sided [-10.84 to 9.15]
Statistical Analysis 2: Comparison: Generic Imiquimod vs Vehicle Cream; Based on Intent-to-Treat Population; Test type: Superiority; p = 0.0001, ANOVA

2. Secondary Outcome: Percentage of Subjects With at Least a 75% Reduction in the Number of AK Lesions From Baseline to End of Treatment (EOT) Visit (Week 16).
Time Frame: Week 16
Population: Using the Intent-to-Treat Population Eighteen (18) ITT subjects from Site 15 are not included due to AK lesion counts not performed post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream
Number analyzed (Participants) | 173 | 171 | 87
Participants | 110 | 114 | 14
Statistical Analysis 1: Comparison: Generic Imiquimod vs Aldara™; Test type: Equivalence — If the 90% confidence interval around the difference between the Generic Imiquimod and Aldara Partial Clearance rates in the PP population were contained within the interval -0.20 to +0.20, then Generic Imiquimod and Aldara were considered to be therapeutically equivalent; Mean Difference (Net) = -3.1, 90% CI 2-sided [-12.11 to 5.95]

3. Secondary Outcome: Percentage of Subjects With at Least a 75% Reduction in the Number of AK Lesions From Baseline to 8 Weeks Post Treatment (Test of Cure Visit).
Time Frame: Week 24
Population: Using Intent-to-Treat population Eighteen (18) ITT subjects from Site 15 are not included due to AK lesion counts not performed post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream
Number analyzed (Participants) | 173 | 171 | 87
Participants | 77 | 77 | 7
Statistical Analysis 1: Comparison: Generic Imiquimod vs Aldara™; Test type: Equivalence — If the 90% confidence interval around the difference between the Generic Imiquimod and Aldara Complete Clearance rates in the ITT population were contained within the interval -0.20 to +0.20, then Generic Imiquimod and Aldara were considered to be therapeutically equivalent; Mean Difference (Net) = -0.5, 90% CI 2-sided [-9.92 to 8.88]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Based on subjects in ITT
Arm/Group | Generic Imiquimod | Aldara™ | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 1/181 | 0/179 | 0/89
Serious Adverse Events (participants affected / at risk) | 4/181 | 2/179 | 2/89
Other Adverse Events (participants affected / at risk) | 79/181 | 60/179 | 25/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Imiquimod (N=181) | Aldara™ (N=179) | Vehicle Cream (N=89)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery atenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Imiquimod (N=181) | Aldara™ (N=179) | Vehicle Cream (N=89)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (7) | 0 (0)
Stomach dicomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Adverse Drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site alopecia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (1)
Hernia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 2 (5) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (7) | 3 (3)
Prostate infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 6 (6) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertrigylceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muskuloskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (7) | 3 (4) | 2 (3)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 3 (4)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 5 (6) | 2 (2)
Lethargy (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Varicose vein ruptured (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.